CLINICAL TRIAL: NCT03452488
Title: Safety and Efficacy of BIO-101 175 mg b.i.d. and 350 mg b.i.d. 26-week Oral Administration to Patients Suffering From Age-related SARcopenia, Including Sarcopenic Obesity, Aged ≥65 Years and at Risk of Mobility Disability
Brief Title: A Double-blind, Placebo-controlled, Randomized INTerventional Clinical Trial (SARA-INT)
Acronym: SARA-INT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biophytis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO101-CL03
Record Dates: First submitted 2018-02-13; First posted 2018-03-02 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sarcopenia; Gait Disorders in Old Age; Muscle Weakness
Keywords: Sarcopenia; Sarcopenic Obesity; 6-minute walking distance; 400 meters walking test; BIO101; Short Physical Performance Battery; Appendicular lean mass
MeSH Terms: conditions — Sarcopenia; Muscle Weakness | interventions — Ecdysterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Each treatment kit showed a preprinted kit number affixed on the primary, secondary and tertiary container. The kit number was assigned via the eCRF after a participant is qualified and was randomized. Neither the Investigator and his staff, nor the Sponsor was aware of the treatment that corresponds to the kit number. The assigned treatment cannot be retrieved from the system, unless a specific unblinding procedure was engaged by the investigator when this was judged necessary by the responsible physician of the investigator center in the context of a severe or serious adverse event.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo was taken orally, two capsules twice daily (BID), 12 hours apart, up to 9 months.
  Interventions: Drug: Placebo
- 175mg BIO101 (Experimental): BIO101 was taken orally, two capsules BID, 12 hours apart, up to 9 months.
  Interventions: Drug: BIO101
- 350mg BIO101 (Experimental): BIO101 was taken orally, two capsules BID, 12 hours apart, up to 9 months.
  Interventions: Drug: BIO101

INTERVENTIONS:
Drug: BIO101 — Oral capsules
  Other Names: 20 hydroxyecdysone (20E)
  Arms: 175mg BIO101; 350mg BIO101
Drug: Placebo — Oral capsules
  Arms: Placebo

SUMMARY:
The main objective of the study is to evaluate the effect of two daily doses of BIO101 versus placebo on mobility function as measured by gait speed using the 400MW test. The absolute change from baseline in meters/second observed in each treatment group at 6 Month was compared to the placebo group. Due to the Covid pandemic >50% of data at endpoint was missing, which may have affected the ability of the study to deliver the expected results. Additionally, although the planned duration of treatment was 6 months, it was extended up to 9 months for some participants as a result of the pandemic.

DETAILED DESCRIPTION:
The aim of this phase 2 double-blind, placebo-controlled, randomized interventional clinical trial (SARA-INT) is to evaluate the safety and efficacy of BIO-101 175 mg b.i.d. and 350 mg b.i.d. 9 months oral administration to participants suffering from age-related sarcopenia, including sarcopenic obesity, aged ≥65 years and at risk of mobility disability. There are 3-arms (2 doses versus placebo). This comparative clinical trial evaluated the effects up to 9 month treatment duration, based on the hypothesis that physical function of sarcopenic, older participants with an initial degree of mobility disability (SPPB) may be improved by BIO101.

Included participants were randomized in a 1:1:1 ratio, to one of the 3 arms of treatment in a blinded manner. The randomization was stratified by gender and by center. Based on absence of long-term toxicology data, the investigational drug exposure was initially capped at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged ≥ 65 years and living in the community, reporting loss of physical function over the last 6-12 months
4. Short Physical Performance Battery (SPPB) score ≤ 8
5. ALM/BMI < 0.789 in men and 0.512 in women, or ALM < 19.75kg in men and <15.02kg in women, as measured by DEXA scan
6. Ability to take oral medication and be willing to adhere to the study intervention regimen.
7. Agreement to adhere to Lifestyle Considerations throughout study duration
8. In the US, women and members of minority groups must be included in accordance with the NIH Policy on Inclusion of Women and Minorities as Participants In Research Involving Human participants.

Exclusion Criteria:

1. Current use of anabolic drugs (e.g. testosterone); current use of Erythropoietin; current use of corticosteroid agents (except local administration route, like eye drops or dermatologic formulations)
2. Non-menopaused women (however ongoing replacement hormonal treatment is not an exclusion criterion)
3. Known allergic reactions to components of the investigational drug.
4. Treatment with another investigational drug or other intervention within three months
5. Unable to understand and perform the functional tests, as judged by the Investigator
6. Inability to perform the 400MW test within 15 minutes
7. Clinical conditions:

   1. Current diagnosis of major psychiatric disorders.
   2. Alcohol abuse or dependence
   3. Severe arthritis
   4. Cancer requiring active treatment (cancer treated with chemotherapy, or radiotherapy and currently on remission is not an exclusion criterion)
   5. Lung disease requiring regular use of supplemental oxygen
   6. Inflammatory conditions requiring regular use of oral or parenteral corticosteroid agents
   7. Severe cardiovascular disease (including New York Heart Association [NYHA] class III or IV congestive heart failure, clinically significant valvular disease, history of cardiac arrest, presence of an implantable defibrillator, or uncontrolled angina)
   8. Parkinson's disease or other progressive neurological disorder
   9. Renal disease requiring dialysis, or known renal insufficiency (moderate or severe reduction in GFR≤30 ml/min/1.73 m2)
   10. Chest pain, severe shortness of breath, or occurrence of other safety concerns during the baseline functional tests 400-meter walk test or 6MWT
   11. History or active signs or symptoms of gallbladder/biliary disease (e.g. previous episodes of cholestasis/biliary tract obstruction, cholelithiasis, cholecystitis, etc.). Of note, history of cholecystectomy and no active biliary signs or symptoms, is not an exclusion criterion.
8. Current physical/rehabilitation therapy (except for passive physical therapy. However, this should not be initiated the week before an evaluation visit and once started, it should be maintained over the study duration).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Van Maanen, Study Director — Biophytis
Locations (22):
- United States (19):
  - Advanced Clinical Research, Banning, California
  - SC Clinical Research, Inc, Garden Grove, California
  - California Research Foundation, San Diego, California
  - Institut On Aging, Gainesville, Florida
  - Jax-Ascent University of Florida, Jacksonville, Florida
  - PANAX Clinical Research, Miami Lakes, Florida
  - Clinical Research of Central Florida, Plant City, Florida
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Jean Mayer USDA Human Nutrition research Center on Aging Tufts University, Boston, Massachusetts
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Columbia University, New York, New York
  - PMJ Research of Wilmington, Wilmington, North Carolina
  - Bowman Gray Center for Medical Education-of- Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Tekton Research, Yukon, Oklahoma
  - Tekton Research, Austin, Texas
  - Medical Center, Houston, Texas
  - Science Advancing Medicine Clinical Research Center, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah
- Belgium (3):
  - Vrije Universiteit Brussel, Brussels
  - Universitaire Ziekenhuizen (UZ) Leuven - Gasthuisberg - Centrum voor metabole botziekten, Leuven
  - Université de Liège, Liège

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 19 centers in the United States and 3 centers in Belgium.
Period: Overall Study
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Started | 81 | 76 | 76
Completed | 70 | 64 | 69
Not Completed | 11 | 12 | 7
Not completed — Adverse Event | 4 | 6 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — PI Decision | 1 | 0 | 0
Not completed — Withdrew consent | 4 | 2 | 2
Not completed — Withdraw due to the COVID-19 outbreak | 1 | 0 | 1
Not completed — Other | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: One participant randomized but not treated with 175 mg BIO101.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101 | Total
Number analyzed (Participants) | 81 | 75 | 76 | 232
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.5 (7.12) | 76.2 (7.10) | 76.3 (6.38) | 76.0 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 37 | 38 | 119
  Male | 37 | 38 | 38 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 13 | 14 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 1 | 11
  White | 65 | 55 | 61 | 181
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 7 | 6 | 7 | 20
  United States | 74 | 69 | 69 | 212

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6 Months in Gait Speed for 400 Meter Walking (MW) Test
Description: Gait speed was measured using the 400 MW test, which measured how long it took the participant to walk a distance of 400 meters. Missing data imputed using adjusted Bayesian Multiple Imputation (MI) methods for Non-Completers who failed to perform the Test feasibility and Multiple Imputation for participants who without data on on-Site visit. Data up to 9 months was used where 6 months data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: Full Analysis Set: The Full Analysis Set (FAS) population consists of randomized participants, excluding participants who failed to take at least one dose of trial medication and had a very early withdrawal (first week after randomization) definitely not related to study medication and lacked any post randomization data. Participants with data available were included.
  One participant randomized but not treated with 175 mg BIO101.
Measure: Least Squares Mean (95% Confidence Interval); unit: Meter/Second (m/s)
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 79 | 75 | 76
Meter/Second (m/s)
  Gait Speed based on Mixed Effect Model: number analyzed (Participants) | 32 | 34 | 40
  Gait Speed based on Mixed Effect Model | 0.0093 [-0.0369 to 0.0556] | 0.0457 [-0.0014 to 0.0927] | 0.0478 [0.0050 to 0.0907]
  Gait Speed Based on Adjusted Bayesian Imputation | -0.2886 [-0.3641 to -0.2132] | -0.2543 [-0.3347 to -0.1738] | -0.2014 [-0.2790 to -0.1238]
  MI + Adjusted Bayesian Imputation | -0.0188 [-0.0743 to 0.0366] | -0.0066 [-0.0547 to 0.0415] | 0.0500 [-0.0013 to 0.1013]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic; Test type: Superiority; p = 0.2437, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic; Test type: Superiority; p = 0.2000, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic based on adjusted Bayesian Imputation; Test type: Superiority; p = 0.3240, Adjusted Bayesian Imputation
Statistical Analysis 4: Comparison: Placebo vs 350mg BIO101; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Gait Speed Based on Adjusted Bayesian Imputation; p = 0.5123, Adjusted Bayesian Imputation
Statistical Analysis 5: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic based on MI and Adjusted Bayesian Imputation; Test type: Superiority; p = 0.6920, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo vs 350mg BIO101; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.0850, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline to 6 Months in Short Form-36 (SF-36) 10 Item Physical Function Domain (PF-10) Sub-score
Description: The Physical Function Domain (PF-10) of the SF-36 assesses an individual's perceived physical functioning and limitations in various activities. It consists of ten items that ask about a person's ability to perform different physical activities and tasks. Scores on the PF-10 range from 0 to 100 where 100 indicates no physical limitations. Missing data imputed using adjusted Bayesian MI methods. Data up to 9 month was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: Full Analysis Set: Population consists of randomized participants, excluding participants who failed to take at least one dose of trial medication and had a very early withdrawal (first week after randomization) definitely not related to study medication and lacked any post randomization data. Participants with data available were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 79 | 75 | 74
score on a scale
  Analysis based on Mixed Effect Model for MMRM: number analyzed (Participants) | 65 | 65 | 68
  Analysis based on Mixed Effect Model for MMRM | 7.3 [2.4 to 12.3] | 7.1 [1.9 to 12.3] | 7.1 [2.2 to 12.1]
  Based on Adjusted Bayesian Imputation | 1.4 [-4.8 to 7.6] | 4.0 [-2.1 to 10.1] | 4.1 [-1.7 to 9.8]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic in Physical Function Domain (PF-10) Sub-score based on Mixed Model Analysis; Test type: Superiority; p = 0.9408, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9485, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic in Physical Function Domain (PF-10) Sub-Score Based on Adjusted Bayesian Imputation; Test type: Superiority; p = 0.9848, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo vs 350mg BIO101; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.5017, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline to 6 Months in Handgrip Strength Test
Description: Handgrip strength was a commonly used measure of upper body skeletal muscle function and had been widely used as a general indicator of frailty with predictive validity for both mortality and functional limitations. Participants were instructed to stand upright and with the dynamometer beside them but not against their body. Strength was measured three times for both hands. The highest value of all 3 attempts was kept for further analysis. Grip strength was measured in the dominant hand using a hydraulic grip strength dynamometer. Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms (Kg)
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 74 | 69 | 69
kilograms (Kg)
  Handgrip strength Test at Month 6 (dominant hand): number analyzed (Participants) | 33 | 33 | 37
  Handgrip strength Test at Month 6 (dominant hand) | -0.709 [-2.902 to 1.484] | -1.601 [-3.935 to 0.733] | 0.590 [-1.533 to 2.712]
  Handgrip strength test at month 6 (Left hand): number analyzed (Participants) | 32 | 32 | 36
  Handgrip strength test at month 6 (Left hand) | -0.860 [-2.852 to 1.131] | -1.597 [-3.766 to 0.573] | 0.319 [-1.626 to 2.264]
  Handgrip strength test at month 6 (Right hand): number analyzed (Participants) | 32 | 34 | 39
  Handgrip strength test at month 6 (Right hand) | -0.842 [-3.098 to 1.414] | -1.664 [-3.993 to 0.665] | 0.865 [-1.262 to 2.992]
  Based on Multiple Imputation (dominant hand) | 0.145 [-2.270 to 2.561] | 0.297 [-2.194 to 2.788] | 0.663 [-1.822 to 3.148]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic in Handgrip Strength Test (dominant hand); Test type: Superiority; p = 0.5200, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3577, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic in Handgrip Strength Test at Month 6 Based on Multiple Imputation (dominant hand); Test type: Superiority; p = 0.9237, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs 350mg BIO101; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.7629, ANCOVA
Statistical Analysis 5: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic in Change from Baseline in Handgrip Strength Test (left hand); Test type: Superiority; p = 0.5695, ANCOVA
Statistical Analysis 6: Comparison: Placebo vs 350mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic in Handgrip Strength Test (Left hand); Test type: Superiority; p = 0.3523, ANCOVA
Statistical Analysis 7: Comparison: Placebo vs 175mg BIO101; Analysis of data collected from baseline to 6 months, or baseline to 9 months due to pandemic in Handgrip Strength Test (Right hand); Test type: Superiority; p = 0.5652, ANCOVA
Statistical Analysis 8: Comparison: Placebo vs 350mg BIO101; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.2472, ANCOVA

4. Secondary Outcome: Change From Baseline to 6 Months in Appendicular Lean Body Mass (ALM) Based on Dual-energy X-ray Absorptiometry (DEXA) Measurements
Description: DEXA scans provided accurate measurements of body composition, recording fat and lean mass distribution throughout the entire body. Foundation of National Health Institute (FNIH) project report recommended ALM alone was used to measure gender-specific low muscle mass. Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Kg
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 58 | 53 | 57
Kg | -0.276 [-0.911 to 0.359] | -0.283 [-0.944 to 0.378] | 0.068 [-0.496 to 0.632]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.9859, ANCOVA — Statistical Analysis of Change from Baseline in ALM
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Statistical Analysis of Change from Baseline in ALM; Test type: Superiority; p = 0.4040, ANCOVA

5. Secondary Outcome: Rate of Response for Completing 400 MW Test After 6 Months
Description: A responder was defined as an improvement (increase) of 0.1 m/s or more in 400MW gait speed test compared to baseline. A non-responder was defined as a participant that was not a responder. Participants with a missing value at the visit and/or missing baseline value were considered as non-responders. Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: Full Analysis Set: Population consists of randomized participants, excluding participants who failed to take at least one dose of trial medication and had a very early withdrawal (first week after randomization) definitely not related to study medication and lacked any post randomization data. Participants with rate of response for completing 400 MW test were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 81 | 75 | 76
Participants
  Responder | 4 | 9 | 11
  Non-responder | 77 | 66 | 65
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.1219, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Test type: Superiority; p = 0.0520, Regression, Logistic

6. Secondary Outcome: Change From Baseline to 6 Months in Muscle Strength Based on Knee Extension
Description: Isometric knee extension torque was measured with a knee extension dynamometer chair. The participants were positioned in an upright position, with straps to affix the hips to the chair and the ankle to a force or torque transducer at the knee angle of 90°. Lever arm length was recorded as the distance between the knee axis of rotation and the middle of the pad. Knee extension was measured using the maximum peak torque measurement Newton meter (Nm) for 60°/s, 90°/s and 180°/s for the tested leg (either right or left). The Knee extension torque was obtained either directly or by multiplying recorded peak force with the lever arm length. The assay with the highest torque output was taken for analyses. Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: Full Analysis Set: Population consists of randomized participants, excluding participants who failed to take at least one dose of trial medication and had a very early withdrawal (first week after randomization) definitely not related to study medication and lacked any post randomization data. This data represents Knee Extension of Highest Reading from all Degrees. Participants with data available were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Newton meter (Nm)
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 8 | 6 | 10
Newton meter (Nm) | 0.484 [-18.088 to 19.056] | -1.092 [-21.833 to 19.649] | -4.515 [-17.889 to 8.858]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.8917, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Test type: Superiority; p = 0.6317, ANCOVA; Mean Difference (Final Values) = -4.999, 95% CI 2-sided [-26.777 to 16.778], Standard Error of Mean 10.2172

7. Secondary Outcome: Change From Baseline to 6 Months in Time for Five Chair Stands as Part of the Short Physical Performance Battery (SPPB) Assessment
Description: The SPPB was a series of tests designed to examine physical movements. The chair stands tests involved standing from a chair a number of times to test leg strength. Each performance measures were assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 the inability to complete the test. The time to complete the task was recorded. The time required to perform five chair stands was scored as follows: ≥ 16.70 sec = 1; 13.70 to 16.69 sec = 2; 11.20 to 13.69 sec = 3; ≤ 11.19 = 4. A score of 0 was assigned to participants unable to perform the task. A summary score ranging from 0 (worst performers) to 12 (best performers) was calculated by adding sub scores from the chair stands test. Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 29 | 31 | 37
Seconds | -3.857 [-6.024 to -1.690] | -2.572 [-4.721 to -0.422] | -1.206 [-3.135 to 0.724]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.3762, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Test type: Superiority; p = 0.0543, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline to 6 Months in Distance in the 6-Minute Walk Test (6MWT)
Description: The 6MWT was a test for functional exercise capacity and involved measuring the distance a participant could cover within the allotted time of 6 minutes. Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 33 | 33 | 37
Meters | -9.879 [-37.089 to 17.330] | -7.166 [-36.559 to 22.228] | 15.728 [-10.981 to 42.436]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.8824, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Test type: Superiority; p = 0.1578, ANCOVA

9. Secondary Outcome: Change From Baseline to 6 Months in Pepper Assessment Tool for Disability (PAT-D) for Obese Participants
Description: The PAT-D was a disability questionnaire which asked respondents how much difficulty they had with a range of activities with functioning. PAT-D scores range from 1 (worst) to 5 (best). Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 38 | 39 | 45
score on a scale | -0.27 [-0.42 to -0.13] | -0.08 [-0.24 to 0.08] | -0.17 [-0.31 to -0.03]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.0511, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Test type: Superiority; p = 0.2771, ANCOVA

10. Secondary Outcome: Change From Baseline to 6 Months in SPPB Total Score
Description: The SPPB was a series of tests designed to examine physical movements. Results of the SPPB included total gait speed score, total balance test score, and total chair stand score. The first tests examined balance (without the assistance of a cane or walker) with the feet in three different orientations, the second test examined gait speed, and the third tests involved standing from a Chair a number of times to test leg strength. A score of 0 was assigned to participants unable to perform the task. A summary score ranging from 0 (worst performers) to 12 (best performers) was calculated by adding sub scores from the walking speed, chair stands and balance tests. Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 56 | 58 | 55
score on a scale | 1.1 [0.5 to 1.6] | 1.00 [0.4 to 1.5] | 0.9 [0.3 to 1.5]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.8084, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Test type: Superiority; p = 0.7266, Mixed Models Analysis

11. Secondary Outcome: Change From Baseline to 6 Months in Sarcopenia Quality of Life (SarQoL) Auto-Evaluation Questionnaire
Description: The SarQoL was a sarcopenia-specific, self-administered, quality of life questionnaire designed for community-dwelling elderly study participants aged 65 years and older.
  The questionnaire contained 22 questions, which took approximately 10 minutes to complete. The questionnaire covered 7 domains: physical and mental health; locomotion; body composition; functionality; activities of daily living; leisure activities; and fears. Most questions are answered on a 4 point Likert scale. The total scoring of the SarQoL questionnaire ranges from 0 (worst imaginable health) to 100 (best imaginable health). A higher score reflected a higher quality of life. Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: Full Analysis Set: Population consists of randomized participants, excluding participants who failed to take at least one dose of trial medication and had a very early withdrawal (first week after randomization) definitely not related to study medication and lacked any post randomization data. This data represents overall disability score. Participants with data available were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 45 | 48 | 51
score on a scale | 8.05 [4.95 to 11.14] | 5.60 [2.43 to 8.78] | 5.83 [2.79 to 8.87]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.2312, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Test type: Superiority; p = 0.2701, Mixed Models Analysis

12. Secondary Outcome: Change From Baseline to 6 Months in Stair Climb Power Test (SCPT)
Description: The SCPT measured the ability to ascend and descend stairs and tests lower body strength and balance and measures time (in seconds) taken to ascend and descend a flight of stairs (10 steps with a 20 cm step height; a handrail was recommended). Step heights should have been suitable (between 16 and 20 cm). Data up to month 9 was used where 6 month data were unavailable for participants enrolled during the COVID-19 pandemic.
Time Frame: Baseline and 6 Months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
Number analyzed (Participants) | 31 | 25 | 34
Seconds | 39.9 [-46.4 to 126.3] | 32.4 [-65.4 to 130.3] | 88.5 [5.1 to 171.8]
Statistical Analysis 1: Comparison: Placebo vs 175mg BIO101; Test type: Superiority; p = 0.8934, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 350mg BIO101; Test type: Superiority; p = 0.3526, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of informed consent until the completion of the study or at the end-of-study visit (up to maximum of 9 months). All ongoing AEs were followed for an additional 30 days after the end-of-study visit.
Description: An AE means any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related (21 CFR 312.32 (a)). Treatment-emergent adverse event (TEAE) is defined as any event that starts on or after the first dose date of study drug up to the last dose date + 6 weeks (date of first randomized study medication intake ≤AE onset date ≥ last dose date + 6 weeks).
Arm/Group | Placebo | 175mg BIO101 | 350mg BIO101
All-Cause Mortality (participants affected / at risk) | 1/81 | 0/75 | 1/74
Serious Adverse Events (participants affected / at risk) | 10/81 | 10/75 | 4/74
Other Adverse Events (participants affected / at risk) | 48/81 | 45/75 | 38/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | 175mg BIO101 (N=75) | 350mg BIO101 (N=74)
AV block third degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic stroke (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Recurrent cardiac decompensation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Unstable angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Calculous cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Partial bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis of leg (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture of intertrochanteric section of femur, closed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer recurrent (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Clot blood (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Ischemic stroke (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
General discomfort (Investigations) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | 175mg BIO101 (N=75) | 350mg BIO101 (N=74)
AV block third degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Age indeterminate inferior myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dizzy on standing (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Increased blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemic stroke (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Recurrent cardiac decompensation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Unstable angina (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vasovagal symptoms (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Deafness temporary (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Persistent postural-perceptual dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Central retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal abrasion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Temporary vision loss (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acid reflux (esophageal) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alternation between constipation and diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bloated feeling (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Calculous cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (2)
Diarrhea recurrent (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
International normalized ratio increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Prothrombin deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Gastro-intestinal disorder NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus of intestine (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2)
Partial bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomited (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (General disorders) | 0 (0) | 1 (1) | 0 (0)
General malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal sores (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (General disorders) | 0 (0) | 1 (1) | 0 (0)
Post fall syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tiredness (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Choledocholithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hemangioma of liver (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic lesion NOS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired liver function (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Steatosis hepatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis of leg (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Common cold (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Flu (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (epidemic) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 3 (3)
Fracture of intertrochanteric section of femur, closed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured nose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration of head (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Low back strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Triglycerides high (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte abnormality (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperamylasemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercholesteremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperlipasemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Worsening of diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Adhesive capsulitis of shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Arthropathy NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Fibula fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flare up of arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fractured toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gait tripping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Myalgia of lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Pain in joint involving forearm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Painful R arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rib pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff tendinitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stiff neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Carcinoma basal cell (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Essential tremor (hereditary) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Foot drop (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Frontal headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Head pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache NOS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Movements disturbance NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor aggravated (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Despondent (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Difficulty sleeping (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Bilateral hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer recurrent (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Creatine kinase increased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cyst of kidney (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Urolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Enlarged prostate (benign) (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute infective bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Bronchitis bacterial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hair growth increased (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hairiness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis suppurativa (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Itchy skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Toe operation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Fall (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Fatigue (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Right cataract extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Wound (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Clot blood (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Hypertension worsened (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension orthostatic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic stroke (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Left deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the coronavirus disease 2019 (COVID-19) outbreak, the implementation of the clinical protocol was affected, including but not limited to the scheduled site visit for safety and/or efficacy, site visits for monitoring, investigational product delivery, collection of adverse events (AEs) and concomitant medications. This led to >50% loss of efficacy data for the primary endpoint and other performance assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT03452488/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03452488/SAP_001.pdf